CLINICAL TRIAL: NCT02566577
Title: Physiologic Effects of RBC Storage in Chronic Transfusion Recipients: Vasoreactivity, Exercise Capacity, and Oxygen Consumption
Brief Title: Physiologic Effects of RBC Transfusion
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulties in recruiting.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Arshed A. Quyyumi, Professor, Emory University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00064523
Record Dates: First submitted 2015-10-01; First posted 2015-10-02 (Estimated); Results first posted 2019-05-24 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Red Blood Cell Transfusion
Keywords: Chronic anemia; Cardiopulmonary testing; Transfusion-dependent anemia
MeSH Terms: interventions — Erythrocyte Count; Blood Transfusion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fresh RBC transfusion/Storage-aged RBC transfusion (Active Comparator): Subjects will receive a transfusion of packed red blood cell (RBC) units of fresh blood (<10 days old) followed by a transfusion of packed RBC units of storage-aged (>21 days old) blood.
  Interventions: Biological: Fresh red blood cell (RBC) transfusion; Biological: Storage-aged red blood cell (RBC) transfusion; Device: Electronic infusion pump
- Storage-aged RBC transfusion/Fresh RBC transfusion (Active Comparator): Subjects will receive a transfusion of packed red blood cell (RBC) units of storage-aged (>21 days old) blood followed by a transfusion of packed RBC units of fresh blood (<10 days old).
  Interventions: Biological: Fresh red blood cell (RBC) transfusion; Biological: Storage-aged red blood cell (RBC) transfusion; Device: Electronic infusion pump

INTERVENTIONS:
Biological: Fresh red blood cell (RBC) transfusion — 1 or 2 cross-matched, packed red blood cells (RBC) units from fresh (<10 days old) blood, as ordered by the attending physician, will be given as an intravenous infusion via a programmable electronic infusion pump (Baxter, Inc) over a period of 1 hour per unit.
Biological: Storage-aged red blood cell (RBC) transfusion — 1 or 2 cross-matched, packed red blood cells (RBC) units from storage-aged (>21 days old) blood, as ordered by the attending physician, will be given as an intravenous infusion via a programmable electronic infusion pump (Baxter, Inc) over a period of 1 hour per unit.
Device: Electronic infusion pump — A programmable, electronic infusion pump (Baxter, Inc) will be used for intravenous transfusion of units of packed red blood cells (RBC). The pump will be programmed to deliver 1 unit of packed RBC per hour.

SUMMARY:
The purpose of this study is to determine how red blood cell transfusions, particularly the length of storage time of units of packed red blood cells, affects the cardiovascular function in patients receiving transfusions. This study will also determine the most ideal way of storing and processing blood, and assess how transfusion affects a person's ability to exercise and how their blood vessels relax and contract.

DETAILED DESCRIPTION:
The purpose of this study is determine red blood cell transfusion, particularly the length of storage time of units of packed red blood cells, affects cardiovascular function in patients receiving transfusions. Transfusion of red blood cells is often used clinically in patients with low red blood cell counts in order to prevent disease progression and death. Recent studies suggest that the use of "aged" versus "fresh" red blood cells is associated with worse clinical outcomes, but there is no clear understanding on how this happens. The investigators want to determine the most ideal way of storing and processing blood, and learn how transfusion affects the ability to exercise in the study subjects and assess the relaxation and contraction of the blood vessels.

ELIGIBILITY:
Inclusion Criteria:

- Subjects with any condition resulting in transfusion-dependent anemia

Exclusion Criteria:

* Age <21 or >80 years
* Pregnancy
* Acute infection in previous 4 weeks
* Active substance abuse within the past year
* Inability to give informed consent
* Inability to return for follow-up
* The presence of alloantibodies that would limit the blood bank's ability to obtain correctly aged red blood cell (RBC) units

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-07; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arshed Quyyumi, MD, FACC, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Radford M, Estcourt LJ, Sirotich E, Pitre T, Britto J, Watson M, Brunskill SJ, Fergusson DA, Doree C, Arnold DM. Restrictive versus liberal red blood cell transfusion strategies for people with haematological malignancies treated with intensive chemotherapy or radiotherapy, or both, with or without haematopoietic stem cell support. Cochrane Database Syst Rev. 2024 May 23;5(5):CD011305. doi: 10.1002/14651858.CD011305.pub3. PMID 38780066

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fresh RBC Transfusion/Storage-aged RBC Transfusion | Storage-aged RBC Transfusion/Fresh RBC Transfusion
Started | 9 | 6
Completed | 6 | 4
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Equipment failure | 1 | 1
Not completed — Physical limitation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fresh RBC Transfusion/Storage-aged RBC Transfusion | Storage-aged RBC Transfusion/Fresh RBC Transfusion | Total
Number analyzed (Participants) | 9 | 6 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 1 | 8
  >=65 years | 2 | 5 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 7 | 4 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 8 | 4 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 6 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Flow-mediated Vasodilation (FMD)
Description: Brachial artery flow-mediated dilation (FMD) will be performed by using ultrasonography. The brachial artery of the non-dominant arm will be imaged using a high-resolution 13 MHz ultrasound transducer. A blood pressure cuff on the forearm will be inflated to supra-systolic pressures to produce 5 minutes of ischemia. After cuff deflation, imaging of the brachial artery will be performed continuously for the next 120 seconds and the flow-mediated dilation will be calculated. Change in FMD is the percent change in the diameter of the brachial artery from baseline (prior to transfusion) to Day 1 (first post-transfusion day). A higher FMD indicates better nitric oxide-dependent endothelial function.
Time Frame: Baseline (prior to transfusion), Day 1 (first post-transfusion day)
Population: The data are not stratified by data points/study periods, as the data points were not collected due to non-compliant nature of the enrolled subjects. Majority of the subjects did not complete the study entirety.
Measure: Mean (Standard Deviation); unit: percentage of FMD
Arm/Group | Fresh RBC Transfusion/Storage-aged RBC Transfusion | Storage-aged RBC Transfusion/Fresh RBC Transfusion
Number analyzed (Participants) | 9 | 6
percentage of FMD | 1.83333 (3.900427) | -3.56667 (6.612614)

2. Primary Outcome: Change in Reactive Hyperemic Index (RHI)
Description: Reactive Hyperemia Index (RHI) will be measured using Pulsatile Arterial Tonometry (PAT). Baseline blood pressure of both hands is measured and PAT probes are placed one on each hand at the same finger (fingers 2, 3 or 4). Following an equilibration period of 10 minutes, the blood pressure cuff will be inflated to 60 mmHg above systolic pressure for 5 minutes followed by deflation of the cuff and the pulsatile recordings from both study and control fingers will be measured. RHI will be calculated from the ratio of the digital pulse volume during reactive hyperemia (following cuff deflation) and baseline. A higher RHI indicates better nitric oxide-dependent endothelial function.
Time Frame: Baseline (prior to transfusion), Day 1 (first post-transfusion day)
Population: Data were not collected. The study subjects could not complete the proposed study procedure due to preexisting comorbidities.
Arm/Group | Fresh RBC Transfusion/Storage-aged RBC Transfusion | Storage-aged RBC Transfusion/Fresh RBC Transfusion
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Maximal Oxygen Uptake (VO2Max)
Description: Subjects will undergo graded treadmill testing following American Heart Association guidelines using the modified Balke protocol. A treadmill with full metabolic cart will be used for the cardiopulmonary testing. Maximal oxygen uptake (VO2Max) is the value achieved when the oxygen uptake remains stable despite a progressive increase in the intensity of exercise. The VO2Max will be calculated from the cardiac output and the arteriovenous oxygen difference during peak exercise. VO2Max is expressed in milliliters of oxygen per minute per kilogram of body weight (ml/min/kg). A higher VO2Max indicates better vascular reactivity.
Time Frame: Day 1 (first post-transfusion day)
Population: as for outcome 2
Arm/Group | Fresh RBC Transfusion/Storage-aged RBC Transfusion | Storage-aged RBC Transfusion/Fresh RBC Transfusion
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Respiratory Exchange Ratio (RER):
Description: Subjects will undergo graded treadmill testing following American Heart Association guidelines using the modified Balke protocol. A treadmill with full metabolic cart will be used for the cardiopulmonary testing. RER is the ratio of VCO2 (carbon dioxide output) to VO2 (oxygen uptake). A higher RER indicates better vascular reactivity.
Time Frame: Day 1 (first post-transfusion day)
Population: as for outcome 2
Arm/Group | Fresh RBC Transfusion/Storage-aged RBC Transfusion | Storage-aged RBC Transfusion/Fresh RBC Transfusion
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: O2 Pulse
Description: Subjects will undergo graded treadmill testing following American Heart Association guidelines using the modified Balke protocol. A treadmill with full metabolic cart will be used for the cardiopulmonary testing. O2 (oxygen) pulse is the amount of O2 consumed from the volume of blood delivered to tissues by each heartbeat; this index is calculated as: O2 pulse = VO2 / heart rate. A higher O2 pulse indicates better vascular reactivity.
Time Frame: Day 1 (first post-transfusion day)
Population: as for outcome 2
Arm/Group | Fresh RBC Transfusion/Storage-aged RBC Transfusion | Storage-aged RBC Transfusion/Fresh RBC Transfusion
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Peak VO2 Lean
Description: Subjects will undergo graded treadmill testing following American Heart Association guidelines using the modified Balke protocol. A treadmill with full metabolic cart will be used for the cardiopulmonary testing. Peak VO2 lean is the peak oxygen uptake adjusted for lean body mass and is reported as a lean body weight-adjustment parameter in mL/kg per minute.
Time Frame: Day 1 (first post-transfusion day)
Population: as for outcome 2
Arm/Group | Fresh RBC Transfusion/Storage-aged RBC Transfusion | Storage-aged RBC Transfusion/Fresh RBC Transfusion
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Oxidative Stress Markers
Description: Oxidative stress will be measured using high-performance liquid chromatography (HPLC) to collect plasma cystine, cysteine, glutathione, and glutathione disulfide levels. Higher levels of cystine, cysteine, glutathione, and glutathione disulfide indicate higher levels of vascular inflammation.
Time Frame: Baseline (prior to transfusion), Day 1 (first post-transfusion day)
Population: as for outcome 2
Arm/Group | Fresh RBC Transfusion/Storage-aged RBC Transfusion | Storage-aged RBC Transfusion/Fresh RBC Transfusion
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change in Levels of Nitric Oxide Metabolites
Description: Nitric oxide metabolites like nitrite, nitrate, S-nitrosothiols (SNO-Hb and SNO-thiol) will be measured from blood samples using high-performance liquid chromatography (HPLC). Higher levels of nitric oxide metabolites indicate higher levels of nitric oxide (NO) synthesis and better vascular reactivity.
Time Frame: Baseline (prior to transfusion), Day 1 (first post-transfusion day)
Population: as for outcome 2
Arm/Group | Fresh RBC Transfusion/Storage-aged RBC Transfusion | Storage-aged RBC Transfusion/Fresh RBC Transfusion
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change in High-sensitivity C-reactive Protein (hsCRP)hsCRP
Description: Levels of high-sensitivity C-reactive protein (hsCRP) in the blood will be measured by using Dade Behring nephelometry. Higher levels of hsCRP indicate increased vascular inflammation.
Time Frame: Baseline (prior to transfusion), Day 1 (first post-transfusion day)
Population: as for outcome 2
Arm/Group | Fresh RBC Transfusion/Storage-aged RBC Transfusion | Storage-aged RBC Transfusion/Fresh RBC Transfusion
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change in Levels of IL-6
Description: Plasma IL-6 concentration will be measured by enzyme-linked immunosorbent assay (ELISA). Change is the difference in the levels of IL-6 from baseline to Day 1 (first post-transfusion day). Higher concentrations of IL-6 indicate increased vascular inflammation.
Time Frame: Baseline (prior to transfusion), Day 1 (first post-transfusion day)
Population: as for outcome 2
Arm/Group | Fresh RBC Transfusion/Storage-aged RBC Transfusion | Storage-aged RBC Transfusion/Fresh RBC Transfusion
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Change in Levels of IL-2
Description: Plasma IL-2 concentration will be measured by enzyme-linked immunosorbent assay (ELISA). Change is the difference in the levels of IL-2 from baseline to Day 1 (first post-transfusion day). Higher concentrations of IL-2 indicate increased vascular inflammation.
Time Frame: Baseline (prior to transfusion), Day 1 (first post-transfusion day)
Population: as for outcome 2
Arm/Group | Fresh RBC Transfusion/Storage-aged RBC Transfusion | Storage-aged RBC Transfusion/Fresh RBC Transfusion
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Four weeks
Arm/Group | Fresh RBC Transfusion/Storage-aged RBC Transfusion | Storage-aged RBC Transfusion/Fresh RBC Transfusion
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/6
Other Adverse Events (participants affected / at risk) | 0/9 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-31): https://cdn.clinicaltrials.gov/large-docs/77/NCT02566577/Prot_SAP_000.pdf